CLINICAL TRIAL: NCT06403722
Title: Perinatal Outcomes in Patients With Suspicion of Preeclampsia and Elevated sFlt-1/PlGF Before Term: A Retrospective Cohort Study
Brief Title: Perinatal Outcomes in Patients With Elevated sFlt-1/PlGF Ratio
Status: Completed | Type: Observational
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Head of the research deparment, Saint Thomas Hospital, Panama
Other Study IDs: 2023-631
Record Dates: First submitted 2024-05-01; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Hypertension in Pregnancy
Keywords: Hypertension, pregnancy induced; Angiogenic factors
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- sFlt-1/PlGF: 110-205: Subjects with suspicion of preeclampsia, with gestational age between 24 - 36 6/7 weeks and sFlt-1/PlGF between 110-205.
  Interventions: Diagnostic Test: Standard of care
- sFlt-1/PlGF: 206-654: Subjects with suspicion of preeclampsia, with gestational age between 24 - 36 6/7 weeks and sFlt-1/PlGF between 206-654.
  Interventions: Diagnostic Test: Standard of care
- sFlt-1/PlGF: 655-999: Subjects with suspicion of preeclampsia, with gestational age between 24 - 36 6/7 weeks and sFlt-1/PlGF between 655-999.
  Interventions: Diagnostic Test: Standard of care
- sFlt-1/PlGF > 1000: Subjects with suspicion of preeclampsia, with gestational age between 24 - 36 6/7 weeks and sFlt-1/PlGF above 1000.
  Interventions: Diagnostic Test: Standard of care

INTERVENTIONS:
Diagnostic Test: Standard of care — No intervention. Clinical evolution was recorded, looking for perinatal complications.

SUMMARY:
Retrospective cohort study that evaluated 190 subjects admitted with diagnosis of hypertensive disorder of pregnancy, between 24 and 36 6/7 weeks, with an sFlt-1/PlGF index greater than or equal to 110. Data were collected on their clinical course prior to termination of pregnancy, using the last reported sFlt-1/PlGF ratio value to classify the population into four cohorts: values between 110-205, between 206 and 654, between 655 and 999 and greater than 1000.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hypertensive disorder of pregnancy
* Gestational age between 24 - 36 6/7
* sFlt-1/PlGF > 110

Exclusion Criteria:

* Gestational age below 23 6/7 weeks and above 37 weeks at the moment of admission.
* Absence of sFLt-1/PlGF ratio result.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects admitted with suspicion of preeclampsia, between 24 and 36 6/7 weeks with result of sFlt-1/PlGF before delivery.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Kidney injury | From the moment of admission up until discharge after delivery, average 5 to 10 days
  Creatinine level > 1.1 Doubling of creatinine levels when others causes had been excluded
Hepatic enzyme abnormalities | From the moment of admission up until discharge after delivery, average 5 to 10 days
  Increase of liver enzyme to > twice the upper limit of normal
HELLP Syndrome | From the moment of admission up until discharge after delivery, average 5 to 10 days
  Elevated liver enzymes Thrombocytopenia Hemolysis
Growth restricted fetus | From the moment of admission up until delivery, average 5 to 10 days
  Fetal weight below 10th percentile and abnormal doppler Fetal weight below 3th percentile
Stillbirth | From the moment of admission up until discharge after delivery, average 5 to 10 days
  Intrauterine fetal demise

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Thomas H, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No